CLINICAL TRIAL: NCT01071174
Title: A Double-Blind, Randomized, Placebo-Controlled Phase I/II Study to Evaluate the Safety of an Intravaginal Matrix Ring With Dapivirine in Healthy, HIV-Negative Women.
Brief Title: A Safety Study of Dapivirine Vaginal Ring in Africa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Annalene Nel, MBChB, PhD, International Partnership for Microbicides
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPM 015
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections
Keywords: HIV infections; Anti-HIV agents; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Ring (Placebo Comparator): Vaginal Ring containing no drug substance
  Interventions: Other: Placebo
- Dapivirine Ring (Experimental): Dapivirine Vaginal Ring 25mg
  Interventions: Other: Dapivirine

INTERVENTIONS:
Other: Dapivirine — Vaginal ring containing 25mg dapivirine; One ring inserted every 28 days for 84 days (3 rings total)
  Arms: Dapivirine Ring
Other: Placebo — Vaginal Ring containing no drug substance
  Arms: Placebo Ring

SUMMARY:
This is a double-blind, randomized, placebo-controlled Phase I/II study to assess the safety of a silicone elastomer vaginal ring containing 25mg dapivirine.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 40 years of age inclusive who can provide informed consent
* Available for all visits and consent to follow all procedures scheduled for the study
* Healthy and self-reported sexually active
* HIV-negative
* On a stable form of contraception and willing to continue OR have undergone surgical sterilization at least 3 months prior to enrollment
* In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle defined as having a minimum of 21 days and a maximum of 35 days between menses
* Upon pelvic/speculum examination and colposcopy at the time of enrolment, the cervix and vagina appear normal as determined by the investigator
* Asymptomatic for genital infections at the time of enrolment
* Willing to refrain from use of vaginal products or objects within 14 days from enrollment and for the duration of the study
* Willing to answer to acceptability, adherence and behavioural assessments throughout the study
* Willing to refrain from participation in any other research study for the duration of their participation
* Willing to provide adequate locator information for study retention purposes and be reachable per local standard procedures

Exclusion Criteria:

* Currently pregnant or last pregnancy within 3 months prior to enrolment
* Currently breast-feeding
* Participated in any other research study within 60 days prior to screening
* Previously participated in any HIV vaccine study
* Untreated urogenital infections within 2 weeks prior to enrolment
* Presence of any abnormal physical finding on the vulva, vaginal walls or cervix during pelvic/speculum examination and/or colposcopy
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, or urethral obstruction, incontinence or urge incontinence
* Pap smear result at screening that requires cryotherapy, biopsy, treatment or further evaluation
* Any Grade 2, 3 or 4 baseline (screening) haematology, chemistry or urinalysis laboratory abnormality according to the DAIDS Table for Grading Adverse Events
* Any abnormal bleeding per vagina, bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrolment
* Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone elastomer
* Any serious acute, chronic or progressive disease
* Any condition(s) that, in the opinion of the investigator, might interfere with adherence to study requirements or evaluation of the study objectives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety as determined by the proportion of women in each arm experiencing protocol-specified events, including AEs, laboratory abnormalities, cervico-vaginal abnormalities, abnormal vaginal flora/pH during the study. | 16 weeks

SECONDARY OUTCOMES:
Acceptability of the product determined by questionnaire. | 16 weeks
Adherence to the protocol-specific product regimen as determined by self-report and clinician observation at each study visit. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Annalene Nel, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (10):
- Kenya Medical Research Institute (KEMRI), Kisumu, Kenya
- University of North Carolina Project, Lilongwe, Malawi
- South Africa (7):
  - Reproductive Health and HIV Research Unit (RHRU), Edendale, KwaZulu-Natal
  - Qhakaza Mbokodo, Ladysmith, KwaZulu-Natal
  - Prevention for HIV and AIDS Project (PHIVA), Pinetown, KwaZulu-Natal
  - Madibeng Centre for Research, Brits, North West
  - Desmond Tutu HIV Foundation Masiphumelele, Cape Town, Western Cape
  - Desmond Tutu HIV Foundation Nyanga, Cape Town, Western Cape
  - Be Part Yoluntu Centre Mbekweni, Paarl, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania

REFERENCES:
- [Derived] Nel A, Bekker LG, Bukusi E, Hellstrӧm E, Kotze P, Louw C, Martinson F, Masenga G, Montgomery E, Ndaba N, van der Straten A, van Niekerk N, Woodsong C. Safety, Acceptability and Adherence of Dapivirine Vaginal Ring in a Microbicide Clinical Trial Conducted in Multiple Countries in Sub-Saharan Africa. PLoS One. 2016 Mar 10;11(3):e0147743. doi: 10.1371/journal.pone.0147743. eCollection 2016. PMID 26963505